CLINICAL TRIAL: NCT02850848
Title: A Randomized, Parallel, Single-Dose Study to Evaluate the Pharmacokinetics of a Test Formulation of Entigin Film Coated Tablet 0.5mg (Entecavir 0.5 mg), Compared to an Equivalent Dose of a Reference Drug Product (Baraclude 0.5mg Tablets) in Healthy Adult Subjects
Brief Title: Pharmacokinetics of Two Formulations of Entecavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YSP RHH3001-01
Record Dates: First submitted 2016-06-16; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis B
Keywords: Pharmacokinetic
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

ARMS (2):
- Entigin Film Coated Tablet 0.5mg (Experimental): Entigin Film Coated Tablet 0.5mg Dosing Regimen: Single dosing of two tablets
  Interventions: Drug: Entigin Film Coated Tablet 0.5mg
- Baraclude 0.5mg Tablets (Active Comparator): Baraclude 0.5mg Tablets Dosing Regimen: Single dosing of two tablets
  Interventions: Drug: (Baraclude 0.5mg Tablets

INTERVENTIONS:
Drug: Entigin Film Coated Tablet 0.5mg
  Arms: Entigin Film Coated Tablet 0.5mg
Drug: (Baraclude 0.5mg Tablets
  Arms: Baraclude 0.5mg Tablets

SUMMARY:
A Randomized, Parallel, Single-Dose Study to Evaluate the Pharmacokinetics of a Test Formulation of Entigin Film Coated Tablet 0.5mg (Entecavir 0.5 mg), Compared to an Equivalent Dose of a Reference Drug Product (Baraclude 0.5mg Tablets) in Healthy

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, aged between 20 to 45 years old.
2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests, chest x-ray and electrocardiogram.

   * no particular clinical significance in clinical examination and laboratory tests within two months (60 days) prior to administration of study medication.
   * normal or considered not clinically significant by the investigator chest X-ray and Electrocardiogram (ECG) results within six months(180 days)prior to administration of study medication.
3. Body weight must be above 50 kg for male and 45 kg for female.
4. The normal range of the body mass index should be between 18 and 30; body mass index equals [weight (kg)]/[height (m)]2.
5. Laboratory determinations results are within normal range or considered not clinically significant by the investigator, including: Serum Glutamic Oxaloacetic Transaminase (SGOT, same as AST), Serum Glutamic Pyruvic Transaminase (SGPT, same as ALT), albumin, glucose, creatinine, uric acid, cholesterol, Triglycerides (TG), Gamma-Glutamyl-Transpeptidase (γ-GT), alkaline phosphatase, total bilirubin, Blood Urea Nitrogen (BUN), Hepatitis B surface antigen (HBsAg), Anti-Hepatitis C virus (HCV) and Anti-Human Immunodeficiency Virus (HIV) test.
6. Hematology test results are within normal range or considered not clinically significant by the investigator, including: hemoglobin, hematocrit, White Blood Cell (WBC) count, Red Blood Cell (RBC) count, platelet count and WBC count with differential.
7. Urinalysis results are within normal range or considered not clinically significant by the investigator, including: glucose, protein, RBC, WBC, epithelial cells, casts and bacteria.
8. Female subject who is:

   * using adequate contraception since last menstruation and no plan for conception during the study.
   * non-lactating.
   * has negative pregnancy test (urine) prior to the study.
9. Informed consent form signed.

Exclusion Criteria:

1. A history of drug or alcohol abuse during the past 24 weeks.
2. Sensitivity to analogous drug.
3. A clinically significant illness (such as lactic acidosis or severe hepatomegaly with steatosis) within the past 4 weeks.
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology within the past 4 weeks.
5. Planned vaccination during the time course of the study.
6. Participation of any clinical investigation during the last 60 days.
7. Regular use of any medication during the last 4 weeks.
8. Single use of any medication during the last 2 weeks.
9. Blood donation of more than 250 mL within the past 12 weeks.
10. Employees and their families of sponsor and/or Contract Research Organization (CRO) company.
11. Individuals are judged by the investigator or co-investigator to be undesirable as subjects.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration(AUC) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr
Time to reach Cmax(Tmax) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr
Peak Drug Concentration(Cmax) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr
Elimination half-life(T1/2) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr
Area under the (first) moment plasma concentration-time curve(AUMC) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr
Mean Residence Time(MRT) | Plasma sample: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 84, 132 and 168 hr Urine sample: -2~0, 0~6, 6~12, 12~24, 24~36, 36~48 hr

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | The safety was monitored throughout the study. Up to 10 weeks